CLINICAL TRIAL: NCT01227642
Title: Phase I/II Evaluation of Cancer-Specific Imaging Using Ultrasound Spectrum Analysis (USA) to Guide Dose Escalated Prostate Brachytherapy
Brief Title: Using Ultrasound Spectrum Analysis (USA) to Guide Dose Escalated Prostate Brachytherapy
Acronym: USA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Collaborators: Riverside Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-147
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Clinical Stage T2b or Less of Prostate Cancer; Prostate Brachytherapy; Transrectal Prostate Ultrasound Treatment Planning
Keywords: Prostate Cancer; Prostate brachytherapy; Ultrasound treatment planning
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pre-implant transrectal ultrasound images and planning (Experimental): Transrectal ultrasound session will be performed at a separate session prior to the implant.
  Interventions: Other: An ultrasound-based technique to identify prostate cancer; Other: pre-implant transrectal ultrasound images and planning; Other: ultrasound-based cancer-specific images

INTERVENTIONS:
Other: An ultrasound-based technique to identify prostate cancer — The technique uses current ultrasound equipment already in use for prostate brachytherapy guidance.By extracting and processing the radiofrequency signal obtained from the ultrasound transducer in ways not done to create the standard B-mode ultrasound image, areas of cancer can be identified and displayed overlying the standard B-mode ultrasound image. Comparing the results with this technique to the results of prostate biopsies demonstrates a high degree of accuracy with the area under the receiver-operator characteristic curve of 0.87, a result superior to any other imaging methods.
Other: pre-implant transrectal ultrasound images and planning — an ultrasound-based technique to identify cancer-containing areas within the prostate.
Other: ultrasound-based cancer-specific images — ultrasound-based cancer-specific images of the prostate prior to the brachytherapy and use them to direct the dosimetry planning
  Other Names: The ultrasound unit used is the B+K Hawk 2102 with probe #8658.

SUMMARY:
In standard treatment, the seeds are placed throughout the prostate to treat the entire prostate. This is done because it was impossible to know where the cancer was located within the prostate. A new technique has been developed using the same ultrasound imaging that you probably had when you had your biopsy. Using this technique, areas likely to contain prostate cancer can be identified.In this early study of 15 subjects, we will test if this method to plan your prostate seed implant is safe and can be done as part of regular care. Areas identified as suspicious for cancer will be treated with higher doses of radiation while those areas not demonstrating cancer will be treated to the standard minimum dose. The higher dose areas will receive two times the minimum dose the prostate usually receives. Because this technique is not perfect, those areas not identified as cancerous should be treated in case there is a cancer area that the technique did not identify. Subjects enrolled in this study will then be followed with this ultrasound technique over the next two years to monitor the changes to the cancerous areas and will undergo a biopsy two years after the procedure. Subjects will, of course, be monitored to assess the success of the technique and its side effects.

DETAILED DESCRIPTION:
Prostate brachytherapy is an increasingly popular treatment for clinically localized prostate cancer.In properly selected patients, it is highly effective with biochemical (PSA) disease free survival rates of 80-87% at 5-10 years.However, the technique is currently limited by the inability to localize the cancer within the prostate. The multifocal nature of prostate cancer is well established. Because of the inability to know where within the prostate the cancer is located, radiation must be delivered throughout the gland. Although this blind approach leads to good results, it is clear that there are regions of the prostate and surrounding tissue that are overexposed to radiation while others are underexposed relative to their true need based on their tumor burden and their proximity to the tumor areas.Feleppa et al. at Riverside Research Institute (New York, NY), a non-profit ultrasound research center, have developed an ultrasound-based technique to identify cancer-containing areas within the prostate. This technique uses current ultrasound equipment already in use for prostate brachytherapy guidance. By extracting and processing the radiofrequency signal obtained from the ultrasound transducer in ways not done to create the standard B-mode ultrasound image, areas of cancer can be identified and displayed overlying the standard B-mode ultrasound image.In this study, we propose to obtain these ultrasound-based cancer-specific images of the prostate prior to the brachytherapy and use them to direct the dosimetry planning.The primary goal of this study is to demonstrate that this imaging modality can be incorporated into the treatment planning process for brachytherapy. Furthermore, we wish to demonstrate the improved dosimetry of the cancer-identified regions while maintaining the urethral dose guidelines noted above. We also wish to compare the differences in dose to the other adjacent normal structures (anterior rectum and right and left neurovascular bundles). Additionally, we seek to demonstrate, at a minimum, no increased toxicity with this approach and similar disease control rates. Of course, ultimately the goal will be to demonstrate a superior therapeutic ratio with this technique.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage ≤ T2b according to the American Joint Commission on Cancer 6th Edition28
* PSA ≤ 10 ng/ml
* Gleason sum on biopsy ≤ 6
* Prostate volume ≤ 50 cc
* Willing to continue follow-up for at least two years.

Exclusion Criteria:

* No prior hormone therapy
* No prior radiotherapy
* No history of collagen vascular disease
* No history of inflammatory bowel disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
modified B+K ultrasound-based tissue-type images | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Ennis, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St.Luke's-Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Result] Ennis RD, Quinn SA, Trichter F, Ryemon S, Jain A, Saigal K, Chandrashekhar S, Romas NA, Feleppa EJ. Phase I/II prospective trial of cancer-specific imaging using ultrasound spectrum analysis tissue-type imaging to guide dose-painting prostate brachytherapy. Brachytherapy. 2015 Nov-Dec;14(6):801-8. doi: 10.1016/j.brachy.2015.06.011. Epub 2015 Jul 31. PMID 26235201